CLINICAL TRIAL: NCT04162275
Title: A Randomized, Double-blind, Placebo-controlled, Single-dose, Dose-escalation Tolerance and Pharmacokinetics Study of Oral Taking Finamine Tablets in Chinese Healthy-adult Subjects
Brief Title: A Single-dose Study to Investigate the Tolerance and Pharmacokinetics of Finamine Tablets in China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yiling Pharmaceutical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: YLCDP-2015-010
Record Dates: First submitted 2019-09-22; First posted 2019-11-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- pre-trial, fasting administration (Experimental): 2 cases were given 150mg Finamine tablets（pre-trial，fasting administration）
  Interventions: Drug: Finamine tablets
- pre-trial,after high fat meal (Experimental): 2 cases were given 150mg Finamine tablets (pre- trial，after high fat meal)
  Interventions: Drug: Finamine tablets
- formal trial-150mg (Placebo Comparator): 4 cases were given 150mg Finamine tablets 2 cases were given placebo
  Interventions: Drug: Finamine tablets; Drug: Placebo tablets
- formal trial-300mg (Placebo Comparator): 6 cases were given 300mg Finamine tablets 2 cases were given placebo
  Interventions: Drug: Finamine tablets; Drug: Placebo tablets
- formal trial-600mg (Placebo Comparator): 6 cases were given 600mg Finamine tablets 2 cases were given placebo
  Interventions: Drug: Finamine tablets; Drug: Placebo tablets
- formal trial-1200mg (Placebo Comparator): 6 cases were given 1200mg Finamine tablets 2 cases were given placebo
  Interventions: Drug: Finamine tablets; Drug: Placebo tablets

INTERVENTIONS:
Drug: Finamine tablets — taken Finamine tablets orally
  Other Names: Finamine tablet
Drug: Placebo tablets — taken Placebo tablets orally
  Arms: formal trial-1200mg; formal trial-150mg; formal trial-300mg; formal trial-600mg

SUMMARY:
Design：Randomization, double-blind, single-center, single-dose, dose-escalation , placebo and parallel control Objectives：

1. To investigate the tolerability and safety of Chinese healthy adult subjects after a single oral administration of Finamine tablets;
2. To investigate the pharmacokinetic (PK) characteristics of Finamine tablets;
3. To provide dose setting basis for follow-up clinical studies. Investigational subject:Healthy-adult subjects in China

34 cases (including 4 cases of the pre- trial), of which the 150mg dose group is in the 4 cases of pre- trial (open, all accepted Finamine tablets orally, among whom, two receive it under fasting condition , and the other two receive it half an hour post a high-fat meal started). There are 6 cases in the formal trial (the subjects' ratio of investigational drug to placebo is 2:1). In all other dose groups, the subjects' ratio of investigational drug to placebo is 3:1.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 65 years old (including the upper and lower limits).
2. Male or female
3. Weight ≥50kg, BMI 18-28 kg/m2 (including the upper and lower limits).
4. Understand and sign the informed consent form，able to understand the process and requirements of the study, and volunteer to participate in this study.

Exclusion Criteria:

If being one of the following conditions, subjects cannot be selected

1. There is a history of disease in heart, liver, kidney, respiratory system, digestive tract, nervous system, endocrine system, immune system, blood system, etc., that the investigator has determined to be clinically significant;
2. Abnormalities are in vital signs, comprehensive physical examinations, laboratory tests, ECG examinations, etc., and they are considered clinically significant by the investigator;
3. Any drug was taken within two weeks prior to dosing in the study , and the investigators believe that this condition may affect the assessment results of this study;
4. There is an seriously allergic history of food and drug or hypersensitivity that the investigator has identified as clinically significant;
5. There are positive results of serological tests (HBsAg, anti-HCV, anti-HIV, or TP-Ab) during screening;
6. Within 1 years prior to the administration of the drug, the history of drinking or drug abuse, that the investigator believes it may affect the evaluation results of the study. Or, during screening, the alcohol breath test or the urine screening test is positive.
7. Subjects cannot quit smoking or quit drinking during the study period or subjects' carbon monoxide breath test is ≥7ppm during the screening period (when the investigator thinks it necessary, it can be further confirmed by urine cotinine test);
8. Subjects participated in any drug clinical trial within 3 months prior to study dosing;
9. Subjects donated blood ≥400mL or 2 units within 3 months prior to study dosing;
10. Subjects do not agree to avoid the use of tobacco ,alcoholic beverages or caffeinated beverages, or to avoid strenuous exercise and other factors that influence such as absorption, distribution, metabolism, and excretion of drugs during 24 hours before dosing in the trial and in the duration of the trial;
11. Pregnant or breastfeeding women, or subjects who are tested positive for serum HCG before dosing in the trial, or who are unable or unwilling to take contraception approved by researchers during the study period as directed by the investigator;
12. Subjects who, in the opinion of nvestigators, are not suitable for participating in this clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Tolerance evaluation | From 0 to 96 hours after dosing
  maximum tolerated dose（MTD）、dose-limiting toxicity（DLT）
AE | From 0 to 96 hours after dosing
  The occurrence rate of AE.
AUC0-96h | From 0 to 96 hours after dosing
  area under the concentration-time curve from the time of dosing extrapolated to the 96h after dosing.
AUCinf | From 0 to 96 hours after dosing
  area under the concentration-time curve from the time of dosing extrapolated to time infinity.
Peak Plasma Concentration (Cmax) | From 0 to 96 hours after dosing
  The PK parameters of the plasma sample.
Tmax | From 0 to 96 hours after dosing
  The amount of time that a drug is present at the maximum concentration in serum.
t1/2 | From 0 to 96 hours after dosing
  The PK parameters of the plasma sample.

CONTACTS AND LOCATIONS:
Locations (1):
- Shijiazhuang Yiling Pharmaceutical Co. Ltd, Shijiazhuang, Hebei, China